CLINICAL TRIAL: NCT01277562
Title: Pilot Study of Secondary Causes of Osteopenia/Osteoporosis in Adults With Breast and Prostate Cancer
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10005
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Prostate Cancer; Osteopenia; Osteoporosis
Keywords: Breast Cancer; Prostate Cancer; Osteopenia; Osteoporosis; Secondary causes of bone loss
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Breast Cancer: Non-metastatic breast cancer with recent diagnosis of osteopenia or osteoporosis
- Prostate Cancer: Non-metastatic prostate cancer with recent diagnosis of osteopenia or osteoporosis

SUMMARY:
The investigators hypothesis is that secondary causes of bone loss are prevalent in patients with breast and prostate cancer, and those patients with secondary causes of bone loss are at higher risk for treatment related bone loss. The goals of this pilot study are to estimate the prevalence of secondary causes of osteoporosis in a cohort of patients with nonmetastatic breast and prostate cancer with osteopenia and osteoporosis.

DETAILED DESCRIPTION:
The interaction of aging, cancer, and bone loss is poorly understood. Cancer or cancer therapy could potentially accelerate bone loss and increase the risk for osteopenia or osteoporosis. The hypothesis of this observational study is that secondary causes of bone loss are prevalent in patients with breast and prostate cancer who are high risk for treatment related bone loss. In order to test this hypothesis, this prospective pilot study will systematically evaluate secondary causes of bone loss in a cohort of patients with nonmetastatic breast and prostate cancer with osteopenia/osteoporosis.

1. Identify patients with nonmetastatic breast cancer newly diagnosed with osteopenia/osteoporosis (Dual Energy X-ray Absorptiometry Bone Density scan T-score average between hip (femoral neck) and spine (L1-L4) of less than -1.0 to -2.5/ less than -2.5, respectively).
2. Identify patients with nonmetastatic prostate cancer newly diagnosed with osteopenia/osteoporosis (Dual Energy X-ray Absorptiometry Bone Density scan T-score average between hip (femoral neck) and spine (L1-L4) of less than -1.0 to -2.5/ less than -2.5, respectively).
3. Refer patient to City of Hope Endocrinology Osteoporosis Clinic.
4. Approach patient in consecutive order in which they have been referred to Endocrinology Osteoporosis Clinic.
5. Describe the study to the patient: patient consents or refuses.
6. Once consented, the patient's medical records are reviewed and Dual Energy X-ray Absorptiometry Bone Density reports are obtained from City of Hope records or the screening medical institution records to confirm diagnosis of osteopenia/osteoporosis or normal bone health.
7. Study participants will undergo an evaluation for secondary causes of bone per standard of care with patient questionnaires.
8. Furthermore, laboratory tests that support secondary causes of bone loss will be retrospectively collected via chart review.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of nonmetastatic breast cancer or diagnosis of nonmetastatic prostate cancer
2. Measurement of bone mineral density by Dual Energy X-ray Absorptiometry (DEXA) within 6 months of enrollment into study.
3. Patients of all ages are eligible but need to qualify for standard DEXA screening
4. Patients of all performance status are eligible
5. Patients are able to give informed consent

Exclusion Criteria

1. Patients previously diagnosed or treated for osteoporosis/osteopenia
2. Stage IV cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with newly diagnosed osteopenia and osteoporosis with diagnosis of non-metastatic breast or prostate cancer
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determine prevalence of secondary causes of bone loss in patients with new diagnosis of osteopenia/o | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arti Hurria, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States